CLINICAL TRIAL: NCT01671189
Title: An Automated SMS-Based Reminder and Rescheduling Tool to Improve Appointment Adherence Rates and Glycemic Control Among Diabetes Patients in San Mateo County
Brief Title: Automated SMS-Based Appointment Validation Tool
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medic Mobile (Industry)
Collaborators: San Mateo Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMMC-MCK-2012
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus Type 2; Adult-onset Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Appointment Reminders (Experimental): 150 patients will be randomly assigned to the intervention arm of the study and receive text reminders about their upcoming appointments.
  Interventions: Other: SMS Reminder Software Tool
- Existing Reminder Protocol (No Intervention): 150 patients will be randomly assigned to the control arm of the study and will not receive SMS reminders about their upcoming appointments. They will, however, be subject to the clinics' existing reminder protocol (phone call reminders by either clinic personnel or computer machine).

INTERVENTIONS:
Other: SMS Reminder Software Tool — The 150 patients in the intervention arm of the study will receive SMS reminders regarding their upcoming appointments. Working in parallel with the SMMC electronic medical records system, the software tool will automate reminders that request text responses from patients to either confirm or request to reschedule their upcoming appointments. This bidirectional text messaging system would not interfere with the clinics' existing reminder protocol.
  Arms: SMS Appointment Reminders

SUMMARY:
Medic Mobile conceptualized and proposed the creation of an SMS-based appointment validation tool to automate appointment confirmation and rescheduling. Working in parallel with the San Mateo Medical Center (SMMC) electronic medical records (EMR) system, the software tool will automate reminders that request text responses from patients to either confirm or request to reschedule their upcoming appointments. While simple in concept, this tool aims to free up scarce clinical resources which are currently allocated to daily patient phone call reminders. With funding from a Bay Area foundation, the investigators will develop and pilot this open-source software tool in a 12-month randomized-controlled trial, slated to begin in October 2012. The endpoints of the study will aim to demonstrate improvements in both appointment adherence and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Belong to Willow Clinic or Fair Oaks Clinic under the San Mateo Medical Center
* Have a diagnosis of type 2 diabetes as indicated by ICD-9 code of 249.xx or 250.xx
* Have a most recent hemoglobin A1c (HbA1c) level greater than 7%
* Are at least 18 years of age
* Have access to cell phone
* Are literate or live with a friend/family member who is literate and willing to handle associated text messages

Exclusion Criteria:

* Have a terminal illness and prognosis of less than one year
* Are unable to demonstrate the ability to reply to an SMS and lack an appropriate proxy
* Are pregnant or expect to be pregnant in the next 6-9 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control (hemoglobin A1c) | 6-9 months post-enrollment
  The hemoglobin A1c (HbA1c) levels of study participants will be measured at the time of enrollment and at the end of the 6-9 month follow-up period.

SECONDARY OUTCOMES:
Appointment Adherence Rate | 6-9 month post-enrollment
  Appointments scheduled during the 6-9 month follow-up period will be systematically tracked and monitored. The proportion of fulfilled appointments will be compared between the intervention and control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Nadim Mahmud, Principal Investigator — Medic Mobile
Locations (1):
- San Mateo Medical Center, San Mateo, California, United States

REFERENCES:
- See also: Medic Mobile — http://www.medicmobile.org